CLINICAL TRIAL: NCT00311220
Title: Phase IV Study of the Quantiferon-RD1 Test
Brief Title: Use TST and QFT-RD1 Test to Monitor the Tuberculous Infection in Patients, Close Contact People and Health Care Workers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); ChungHwa Veterans house (Unknown); Taiwan Province Tau-Wein Hospital (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TCVGH-940117/439
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2006-04

CONDITIONS: Tuberculosis; Latent Tuberculosis; Tuberculosis Contact; Elderly
Keywords: tuberculosis; latent tuberculosis; tuberculin skin test; quantiferon TB-RD1; contact screening; elderly
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Tuberculin; Skin Tests

INTERVENTIONS:
Drug: tuberculin for skin test

SUMMARY:
Tuberculosis is still the most common infectious disease in Taiwan. The infants in Taiwan have been vaccinated at birth with BCG -Tokyo 171 strain since 1951. The BCG vaccination rate is 97% among first grade students in a recent national survey. Even with such a high BCG vaccination coverage, Taiwan still has a relatively high TB incidence rate. In 2004, there were totally 16,784 newly diagnosed TB cases and the annual incidence was 74.11 per 100,000 population nationally. Nearly 70% of the incidence cases were men and 30.4% were women. The mean age of incidence cases was 57.8 years old (median=63). 8,440(50.29%) patients were elderly than 65 years old. The elderly men did not receive the BCG vaccination and were the most important group to develop newly diagnosed tuberculosis and a special issue for the national TB control program in Taiwan.

The tuberculin skin test (TST) is the only widely available method for detecting whether people have an immunologic reactivity to mycobacterial antigens and identified as latent tuberculosis infection (LTBI). Targeted tuberculin testing for latent TB infection is a very important strategy to identify subjects with high risk to develop tuberculosis including those who have recent infection with Mycobacterium tuberculosis or have clinical conditions that associated with an increased risk for progression of LTBI to active TB but the sensitivity was lower in elderly patients.

Quantiferon-TB gold test (QFT-RD1) is a new diagnostic test for latent tuberculosis and a valuable alternative to skin testing. This whole-blood assay measures the production of IFN-  in whole blood upon stimulation by ESAT-6 and CFP-10 and allows distinction of latent M. tuberculosis infection from BCG-induced reactivity. ESAT-6 and CFP-10 are deleted from BCG Region 1 (RD1), not present in most nontuberculous mycobacteria and are highly specific indicators of M. tuberculosis infection. Thus, the aim of this study was to estimate the specificity and sensitivity of a whole blood IFN-γassay employing CFP-10 and ESAT-6, for the detection of M. tuberculosis infection in a clustered high risk elderly population.

Changhwa Veterans Home is a government-expense veterans home with totally 519 residents in 2004.The inhabitants were all elderly people and lived in groups. , They did not receive BCG vaccination and were the high risk group to develop endemic TB infection. The annual TB incidence rate over there was 3,500 per 100,000 population.

DETAILED DESCRIPTION:
STUDY POPULATION AND METHODS Population The study population represented individuals screened for TB over a 6-month period ending in December 2004 as part of a number of community health outreach programs based at the Center of Disease Control in Taichung, Taiwan. Changhwa Veterans Home is a government-expense veterans home with totally 519 residents in 2004. Only individuals with a properly read TST and signed informed consent were included in the study population. If a TST was positive, further evaluation for TB was advised. Anyone found to have active TB infection (12 individuals diagnosed, all from household contacts) was appropriately treated and were also included from the study. No general population low-risk controls were included in the study population. There were no other entry exclusions for the study. Before the TST was administered, a short interview including verbal consent and a BCG scar count evaluation was conducted by an experienced nurse.

The TST contained 2 tuberculin units (TU) of RT23 tuberculin with Tween 80 (0.2 ml of 1TU/0.1 ml) given intradermally on the left forearm volar surface by Mantoux technique. Validity measures such as inter-observer performance were done for TST placement or interpretation individually by two experienced nurse. A purified protein derivative-Siebert (PPD-S) dose of 5TU is roughly equivalent to the 2TU of RT23. 2TU is the International Union Against Tuberculosis and Lung Disease recommended dose for RT23 TST. TST was also performed on BCG-vaccinated health care workers . After 48-72 h of injection, the TST site should be evaluated for induration and a transverse measurement was recorded. Any readings made outside of the above time period were excluded from the study. All unvaccinated subjects had their blood drawn for the QFT-RD1 the same time with applying the first TST. A TST reaction size of ≧10 mm was interpreted as a 'positive' TST which guided any further medical evaluation. This is the traditional cutoff point used for RT23 tuberculin in Taiwan as well as in most studies worldwide. If initial TST diameter less than 10 mm, second TST was repeated within 1-5 weeks to observe any 'boosting phenomenon' was possible. Statistical analysis of skin test results for each population characteristic was done at this cut-off point, with the exception of one analysis specifically done at≧18 mm in BCG-vaccinated health care workers.

Household contacts of active TB patients were presumably at highest risk for TB infection; the group was labeled 'household contact'. No active TB cases have been reported among these residents for years.

ELIGIBILITY:
Inclusion Criteria:

* people close contact with active tuberculosis patients including health care workers, people in the veterans home, and/or the close contact family or high risk area or county
* low risk volunteers : the clerk and interns doctors initially in the hospital training

Exclusion Criteria:

* HIV

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2004-01; Study Completion 2006-11

PRIMARY OUTCOMES:
tuberculin skin test positive rate
quantiferon positive rate

SECONDARY OUTCOMES:
two steps tuberculin skin test
active tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Shen Gwan Han, MD, Principal Investigator — Division of Chest Medicine, Department of Internal Medicine, Taichung Veterans General Hospital
Locations (1):
- Division of Chest Medicine, Department of Internal Medicine, Taichung Veterans General Hospital, Taichung, Taiwan, China